CLINICAL TRIAL: NCT02933866
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel-Design, Multiple-Site, Phase III Clinical Study to Evaluate the Efficacy and Safety of DSXS Topical Product in Patients With Mild to Severe Scalp Psoriasis
Brief Title: Phase III Clinical Study in Patients With Mild to Severe Scalp Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSXS 1536
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Scalp Psoriasis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DSXS topical (Experimental): applied once daily for 28 days
  Interventions: Drug: DSXS topical
- Vehicle topical (Placebo Comparator): applied once daily for 28 days
  Interventions: Drug: Vehicle topical

INTERVENTIONS:
Drug: DSXS topical — topical treatment
  Other Names: Active
  Arms: DSXS topical
Drug: Vehicle topical — topical treatment
  Other Names: placebo
  Arms: Vehicle topical

SUMMARY:
A Randomized, Double-Blind, Vehicle-Controlled, Parallel-Design, Multiple-Site, Phase III Clinical Study to Evaluate the Efficacy and Safety of DSXS topical product in Patients with Mild to Severe Scalp Psoriasis

DETAILED DESCRIPTION:
To evaluate the therapeutic efficacy and safety of DSXS topical product (Taro Pharmaceuticals, U.S.A., Inc.) compared to a Vehicle topical product (Taro Pharmaceuticals, U.S.A., Inc.) in patients with mild to severe scalp psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females 18 years of age and older.

Exclusion Criteria:

* Females who are pregnant, lactating or likely to become pregnant during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novum Pharmaceutical Research Services, Study Chair — http://www.novumprs.com/contact
Locations (1):
- Taro Pharmaceuticals USA, Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DSXS Topical | Vehicle Topical
Started | 186 | 185
Completed | 174 | 176
Not Completed | 12 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DSXS Topical | Vehicle Topical | Total
Number analyzed (Participants) | 186 | 184 | 370
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (15.9) | 49.3 (16.7) | 50.1 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 111 | 219
  Male | 78 | 73 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 84 | 83 | 167
  Not Hispanic or Latino | 102 | 101 | 203
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 7 | 11 | 18
  White | 171 | 167 | 338
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 186 | 184 | 370
Percent Scalp Affected [Mean (Standard Deviation); unit: percent] | 33.7 (26.0) | 29.2 (23.8) | 31.4 (25.0)
Number of months and/or years patient has suffered from symptoms caused by scalp psoriasis [Count of Participants; unit: Participants]
  <= 3 Months | 18 | 19 | 37
  > 3 Months And <= 6 Months | 1 | 3 | 4
  > 6 Months And <= 1 Year | 8 | 6 | 14
  > 1 Year And <= 3 Years | 38 | 33 | 71
  > 3 Years And <= 5 Years | 19 | 31 | 50
  > 5 Years | 102 | 92 | 194

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients in Each Treatment Group Who Are Considered a Clinical Success
Description: Clinical Success is defined by an IGA score of 0 (clear) or I (almost clear) with at least a 2 grades reduction from baseline at Day 29 ± 2
Time Frame: Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS Topical | Vehicle Topical
Number analyzed (Participants) | 186 | 184
Participants | 49 | 41
Statistical Analysis 1: Comparison: DSXS Topical vs Vehicle Topical; Test type: Superiority; p = 0.2961, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | DSXS Topical | Vehicle Topical
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/183
Serious Adverse Events (participants affected / at risk) | 0/183 | 0/183
Other Adverse Events (participants affected / at risk) | 31/183 | 42/183
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSXS Topical (N=183) | Vehicle Topical (N=183)
Application site dermatitis (General disorders) | 1 (1) | 0 (0)
Application site dryness (General disorders) | 2 (2) | 1 (2)
Application site exfoliation (General disorders) | 1 (1) | 0 (0)
Application site hyperaesthesia (General disorders) | 0 (0) | 1 (1)
Application site irritation (General disorders) | 1 (1) | 0 (0)
Application site pain (General disorders) | 2 (2) | 6 (6)
Application site paraesthesia (General disorders) | 0 (0) | 1 (3)
Application site pruritus (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 7 (8) | 9 (11)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 4 (4) | 11 (13)
Eye pain (Eye disorders) | 0 (0) | 4 (4)
Ocular hyperaemia (Eye disorders) | 2 (2) | 1 (1)
Ocular icterus (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-06-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT02933866/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT02933866/SAP_001.pdf